CLINICAL TRIAL: NCT06597864
Title: Seven-step Phenomenological Psychotherapy for Self-disorder - a Pilot Study
Acronym: SSPP-SD-p
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Tor Gunnar Værnes, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 750920
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Psychosis;Schizophrenic
Keywords: self-disorder; psychotherapy; phenomenology; qualitative; schizophrenia spectrum; psychosis risk syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy group (Other): Single arm of participants receiving a phenomenologically oriented psychotherapeutic intervention
  Interventions: Behavioral: Seven-step phenomenological psychotherapy for self-disorders

INTERVENTIONS:
Behavioral: Seven-step phenomenological psychotherapy for self-disorders — Phenomenological exploration of anomalous self-experiences, meaning attributions and behavioral consequences. Psychoeducation. Dialogical approach focusing on self-narratives, searching for new meaning and understanding of self-disorders

SUMMARY:
The goal of this clinical pilot study is to learn how adults with schizophrenia or other non-affective psychotic disorders or psychosis risk syndromes experience a novel psychotherapeutic treatment for self-disorders. The study has a qualitative, phenomenological research design. After end of treatment, the participants are interviewed about the experience of the treatment. This include how the participants liked it, if it was experienced as helpful and useful, and changes in self-experience and experience of relations to others and the world.

DETAILED DESCRIPTION:
Self-disorders are considered as central features of schizophrenia spectrum disorders which may be present both before, during, and after psychotic episodes. They are characterized by disturbances in the sense of ownership to experiences and agency of action, as well as in the sense of presence, reality and existence. They are further considered to drive symptom development during prodromal schizphrenia. Self-disorders may be very painful, and associated with anxiety, disturbances in daily functioning and increased sucidality. There is a lack of studies investigating the effect of psychotherapy on self-disorders. Hence, there is a need for developing and testing new treatment approaches to these debilitating conditions.

In this pilot study the investigators want to test a new model and manual for the treatment of self-disorders, the Seven-Step Phenomenological Psychotherapy for Self-Disorder (SSPP-SD), first developed by Dr.Med Paul Møller. This model focuses on the phenomenological exploration of self-disorders, subjective understanding, meaning and associated behaviors, psychoeducation, and the joint exploration of new meanings and understanding related to the experiences. The length of the treatment is stipulated to 14 individual sessions over 7-10 weeks. The first step of the treatment involves a semi-structured interview with the Examination of Anomalous Self-Experience (EASE).

The study has a qualitative phenomenological design where the primary research question is how the participants experienced the treatment. In more detail, the investigators want to explore both positive and negative experiences, how useful or helpful the participants experienced the treatment, and how the treatment affected self-experience and experience of relations to others and the world. These experiences will be explored in a qualitative interview following the end of treatment. In addition, the participants will answer questionnaires regarding symptoms, functioning, life quality (before and after treatment) and satisfaction with the treatment (after treatment). The study will inform the planning of a larger clinical trial testing the effect of the SSPP-SD on self-disorders in participants with psychotic disorders at Vestre Viken Hospital, Norway. Hence, in this pilot study the investigators will also register and evaluate therapist experiences of the SSPP-SD, and fidelity to the manual. The therapists will be supervised by Dr.med Paul Møller.

Six participants with schizophrenia or other ICD-10 F20-29 disorders, or with psychosis risk syndromes as defined in the Structured Interview for Psychosis-risk Syndromes (SIPS) will be included. They will be included from an outpatient clinic for psychotic disorders at Akershus University Hospital, Norway. Two experienced therapists trained in the model will offer the therapy, including project leader Dr. Tor Gunnar Værnes at the Oslo University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses in the ICD-10-CM Code range, i.e. schizophrenia, schizotypal, delusional, and other non-mood psychotic disorders. First diagnosed no more than 3 years ago.
* Or Psychosis risk syndrome as defined in the Structured Interview of Psychosis-Risk Syndromes (SIPS) (McGlashan, Walsh, & Woods, 2010)
* Present with anomalous self-experiences, as confirmed by the Screen Questionnaire for EASE (SQuEASE-6) (Møller, 2018)
* Motivated to explore and work with anomalous self-experiences in psychotherapy

Exclusion Criteria:

* Severe, ongoing psychosis
* Severe, ongoing drug abuse
* IQ<70
* Poor Norwegian language profiency

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Experience of the seven-step phenomenological psychotherapy model for self-disorders | After completing the SSPP-SD treatment, up to 12 weeks after study inclusion
  Qualitative, semi-structured interview exploring how the participants experienced the therapy.

SECONDARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Self-report of anxiety symptoms scored on a 0-3 Likert scale. Min-max score on the total scale: 0-21. Higher scores reflect more severe symptoms/outcome
Patient Health Questionnaire-9 (PHQ-9) | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Self-report of 9 depression symptoms. Each symptom scored on a 0-3 Likert scale. Min-max scores 0-27. Higher scores imply a more severe outcome
Work and Social Adjustment Scale (WSAS) | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Self-report measure for impairment in social and work functioning and adjustment. It includes 5 items to be scored on a 0-8 Likert scale. Min-max score 0-40. Higher scores imply a more severe outcome
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Self-report measure for mental well-being. It includes 14 items each scored on a 1-5 Likert scale. Min-max score: 14-70. Higher scores imply a more severe outcome.
Positive and Negative Syndrome Scale-6 (PANSS-6) | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Brief rating scale for the measurement of severity in schizophrenia. A semi-structured interview assessing 3 positive and 3 negative symptoms. Each symptom scored on a 1-7 Likert scale. Min-max total score: 6-42. Higher scores imply more severe outcomes
10-point self-disorder questionnaire | Before the SSPP-SD intervention and at the end of the intervention, up to 12 weeks after enrollment
  Brief rating scale for the measurement of self-disorders. It includes 10 items, each scored on a 0-4 Likert scale. Min-max score 0-40. Higher scores imply a more severe outcome
Examination of Anomalous Self-Experience (EASE) | During the first of sevens steps of treatment, session 1 and 2. Up to 3 weeks after study enrollment
  Semi-structured interview for a qualitative exploration and quantitative assessment of anomalous self-experiences. It includes 57 main items, each scored on a 0-4 Likert scale (it also include a range of subitems which are scored on a 0-4 Likert scale, but the scores on these subitems are not included in the total EASE score). Min-max total score 0-228. Higher scores imply more severe outcomes
Client Satisfaction Questionnaire (CSQ-8) | After end of SSPP-SD treatment, up to 12 weeks after enrollment
  Self-report measure of satisfaction with health-care, including 5 questions. Each question scored on a 0-4 Likert scale. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Gunnar Værnes, Dr.philos., Principal Investigator — Oslo University Hospital, Early Intervention in Psychosis Advisory Unit for South-East Norway
Locations (2):
- Norway (2):
  - Bærum DPS, Sandvika, Bærum
  - Akershus University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
Due to the qualitative, phenomenological design, and the small number of participants